CLINICAL TRIAL: NCT02380274
Title: A Prospective Observational Cohort Study of Patients With Castration-Resistant Prostate Cancer (CRPC) in the United States
Brief Title: Observational Cohort Study of Patients With Castration-Resistant Prostate Cancer (CRPC)
Acronym: TRUMPET
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: ONC-MA-1004
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer; Metastatic Prostate Cancer
Keywords: Prostate Cancer; Castration-resistant Prostate Cancer; Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CRPC: Patients with CRPC

SUMMARY:
The purpose of this study is to describe patterns of care in CRPC patients, as well as health-related quality of life (HRQoL) outcomes associated with CRPC and its management.

This study will also describe factors influencing treatment decisions including reason(s) for treatment choices and triggers for treatment changes for CRPC as well as describe clinical outcomes based on patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion:

* Patient may have M0 or M1 disease
* Confirmed diagnosis of CRPC defined by both Testosterone at castrate levels, as evidenced by a serum testosterone level ≤ 1.73 nmol/L (50 ng/dL) and Clear progressive disease, as evidenced by a minimum of two rising PSA levels measured at least 7 days apart or new clinical or imaging evidence of progressive metastatic disease
* Initiating the first or second line treatment for CRPC: including anti- androgens, androgen synthesis inhibitors, chemotherapy, immunotherapy or radionuclide therapy. Previous first line CRPC treatments are limited to: First generation anti-androgens (bicalutamide, flutamide, or nilutamide) or Sipuleucel-T
* Patients may be enrolled within 90 days from the time of decision to treat or within 90 days of treatment initiation.
* Willing and able to complete periodic patient-reported outcome (PRO) questionnaires, with or without assistance
* Estimated life expectancy of ≥ 6 months

Caregiver Inclusion:

* Meets the definition of an unpaid relative or friend who helps the patient with his or her activities of daily living
* Willing and able to complete caregiver-reported outcome questionnaires over the course of the patient's participation in the study

Exclusion Criteria:

Patient Exclusion:

* Receiving concomitant treatment for other cancer (excluding basal cell carcinoma, squamous cell carcinoma and treatment for hormone sensitive prostate cancer) within 6 months prior to enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male patients diagnosed with CRPC. Eligible patients will be enrolled by urologists and medical oncologists.
Sampling Method: Non-Probability Sample
Enrollment: 1030 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Number of CRPC Treatment Patterns | Up to 6 years following enrollment onto the study
  Treatment patterns will be described according to: The distribution and timing of disease assessment methods (PSA, other laboratory testing, imaging); Treatment settings; Physician referral patterns from urologist to oncologist (occurrence and timing of referrals) where applicable; CRPC treatments, including initial choices, sequencing and entry into interventional clinical trials
Health-related Quality of Life (HRQoL) as assessed by Modified Total Illness Burden Index (TIBI-CaP) | Baseline
HRQoL as assessed by SF-12v2 Health Survey | Baseline and up to 6 years approximately every 3 months
HRQoL as assessed by Functional Assessment of Cancer Therapy-Prostate (FACT-P) | Baseline and up to 6 years approximately every 3-6 months
HRQoL as assessed by Brief Pain Inventory - Short Form (BPI-SF) | Baseline and up to 6 years approximately every 3 months
HRQoL as assessed by Memorial Anxiety Scale for Prostate Cancer (MAX-PC) | Baseline and up to 6 years approximately every 3 months
HRQoL as assessed by Work Productivity and Activity Questionnaire: Specific Health Problem (WPAI-SHP) | Baseline and up to 6 years approximately every 3-6 months
HRQoL as assessed by Service Satisfaction Scale for Cancer Care (SCA) | Baseline and up to 6 years approximately every 3-6 months

SECONDARY OUTCOMES:
Number of patients with Physician Factors for Treatment Decisions | Up to 6 years following enrollment onto the study
  Physician-reported primary factor in treatment decision making and identified trigger for change will be categorized as:Progressive disease (by Prostate specific antigen (PSA), radiographic, or other unequivocal clinical progression); Tolerability (Lack of tolerability or intolerable side effects); Availability of investigational product/clinical trial; Specific patient concerns regarding treatment; Insurance coverage/costs; Patient compliance
Number of patients with Clinical outcomes, including PSA values, clinical and/or radiologic evidence of disease progression and overall survival | Up to 6 years following enrollment onto the study
Number of patients with Prognostic factors (e.g., patient and disease characteristics) potentially related to select clinical outcomes and HRQoL | Up to 6 years following enrollment onto the study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — APGD, Medical Affairs, Americas
Locations (148):
- United States (148):
  - Site USSUB1007, Homewood, Alabama
  - Site USSUB1010, Anchorage, Alaska
  - Site USSUB1111, Phoenix, Arizona
  - Site US1104, Scottsdale, Arizona
  - Site US1065, Tucson, Arizona
  - Site USSUB1033, Tucson, Arizona
  - Site US1121, Yuma, Arizona
  - Site US1198, Hot Springs, Arkansas
  - Site US1229, Fresno, California
  - Site US1093, Highland, California
  - Site US1085, Laguna Hills, California
  - Site US1087, Los Angeles, California
  - Site USSUB1038, Marina del Rey, California
  - Site US1167, Sacramento, California
  - Site USSUB1026, San Diego, California
  - Site US1089, San Diego, California
  - Site USSUB1037, San Jose, California
  - Site US1148, Santa Monica, California
  - Site USSUB1099, Templeton, California
  - Site US1055, Torrance, California
  - Site USSUB1001, Denver, Colorado
  - Site US1032, Englewood, Colorado
  - Site US1147, Glenwood Springs, Colorado
  - Site US1086, Norwich, Connecticut
  - Site US1160, Stamford, Connecticut
  - Site US1205, Bay Pines, Florida
  - Site USSUB1014, Daytona Beach, Florida
  - Site US1129, Fort Lauderdale, Florida
  - Site US1101, Fort Myers, Florida
  - Site US1073, Hialeah, Florida
  - Site US1102, Lakewood Rch, Florida
  - Site US1105, Naples, Florida
  - Site US1108, Naples, Florida
  - Site US1067, Albany, Georgia
  - Site USSUB1025, Atlanta, Georgia
  - Site US1051, Newnan, Georgia
  - Site US1172, Thomasville, Georgia
  - Site US1066, Boise, Idaho
  - Site USSUB1018, Coeur d'Alene, Idaho
  - Site US1090, Chicago, Illinois
  - Site US1184, Crystal Lake, Illinois
  - Site US1084, Glenview, Illinois
  - Site US1213, Hines, Illinois
  - Site US1204, North Chicago, Illinois
  - Site US1119, Urbana, Illinois
  - Site USSUB1035, Greenwood, Indiana
  - Site USSUB1009, Jeffersonville, Indiana
  - Site US1201, Lafayette, Indiana
  - Site US1203, Davenport, Iowa
  - Site USSUB1072, Wichita, Kansas
  - Site US1079, Wichita, Kansas
  - Site US1139, Ashland, Kentucky
  - Site USSUB1049, Baton Rouge, Louisiana
  - Site US1181, Covington, Louisiana
  - Site US1164, Houma, Louisiana
  - Site US1061, New Orleans, Louisiana
  - Site US1115, New Orleans, Louisiana
  - Site US1004, Shreveport, Louisiana
  - Site US1118, Lewiston, Maine
  - Site US1052, Bethesda, Maryland
  - Site US1133, Greenbelt, Maryland
  - Site USSUB1042, Towson, Maryland
  - Site US1077, Worcester, Massachusetts
  - Site US1039, Worcester, Massachusetts
  - Site US1233, Detroit, Michigan
  - Site US1187, Lansing, Michigan
  - Site US1056, Royal Oak, Michigan
  - Site USSUB1143, Troy, Michigan
  - Site US1174, Duluth, Minnesota
  - Site US1157, Minneapolis, Minnesota
  - Site USSUB1063, Saint Cloud, Minnesota
  - Site US1151, Saint Louis Park, Minnesota
  - Site US1120, Woodbury, Minnesota
  - Site US1080, Tupelo, Mississippi
  - Site US1144, Bolivar, Missouri
  - Site US1081, Columbia, Missouri
  - Site US1223, St Louis, Missouri
  - Site US1123, Billings, Montana
  - Site USSUB1062, Billings, Montana
  - Site USSUB1048, Missoula, Montana
  - Site US1070, Fremont, Nebraska
  - Site US1165, Grand Island, Nebraska
  - Site US1149, Omaha, Nebraska
  - Site USSUB1022, Omaha, Nebraska
  - Site US1166, Belleville, New Jersey
  - Site US1169, Berkeley Heights, New Jersey
  - Site US1059, Edison, New Jersey
  - Site USSUB1006, Englewood, New Jersey
  - Site US1156, Paramus, New Jersey
  - Site USSUB1016, Voorhees Township, New Jersey
  - Site US1053, Albuquerque, New Mexico
  - Site US1189, Santa Fe, New Mexico
  - Site USSUB1041, Albany, New York
  - Site US1226, Buffalo, New York
  - Site US1142, Cheektowaga, New York
  - Site USSUB1023, East Setauket, New York
  - Site US1127, Garden City, New York
  - Site US1163, Jamaica, New York
  - Site US1071, Manhattan, New York
  - Site US1046, Mineola, New York
  - Site US1054, North Hills, New York
  - Site USSUB1012, Poughkeepsie, New York
  - Site USSUB1043, Syracuse, New York
  - Site US1068, The Bronx, New York
  - Site US1044, Asheville, North Carolina
  - Site US1064, Concord, North Carolina
  - Site US1132, Durham, North Carolina
  - Site US1136, Gastonia, North Carolina
  - Site USSUB1017, Greenville, North Carolina
  - Site USSUB1134, Hendersonville, North Carolina
  - Site US1069, High Point, North Carolina
  - Site US1030, Pinehurst, North Carolina
  - Site USSUB1036, Raleigh, North Carolina
  - Site US1078, Washington, North Carolina
  - Site US1074, Winston-Salem, North Carolina
  - Site US1141, Winston-Salem, North Carolina
  - Site USSUB1011, Cincinnati, Ohio
  - Site USSUB1028, Middleburg Heights, Ohio
  - Site USSUB1058, Oklahoma City, Oklahoma
  - Site US1137, Oklahoma City, Oklahoma
  - Site US1153, Coos Bay, Oregon
  - Site US1116, Corvallis, Oregon
  - Site US1230, Portland, Oregon
  - Site USSUB1020, Springfield, Oregon
  - Site USSUB1003, Bala-Cynwyd, Pennsylvania
  - Site US1100, Lancaster, Pennsylvania
  - Site US1218, Pittsburgh, Pennsylvania
  - Site US1224, Charleston, South Carolina
  - Site USSUB1002, Myrtle Beach, South Carolina
  - Site USSUB1095, Watertown, South Dakota
  - Site USSUB1031, Chattanooga, Tennessee
  - Site US1024, Cookeville, Tennessee
  - Site US1128, Nashville, Tennessee
  - Site US1131, Nashville, Tennessee
  - Site USSUB1088, Nashville, Tennessee
  - Site US1227, Dallas, Texas
  - Site US1140, Fort Worth, Texas
  - Site US1208, San Antonio, Texas
  - Site USSUB1045, Temple, Texas
  - Site US1207, Salt Lake City, Utah
  - Site US1092, Richmond, Virginia
  - Site US1096, Richmond, Virginia
  - Site USSUB1005, Virginia Beach, Virginia
  - Site US1083, Bellingham, Washington
  - Site US1029, Everett, Washington
  - Site US1112, Tacoma, Washington
  - Site US1122, La Crosse, Wisconsin
  - Site US1232, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.